CLINICAL TRIAL: NCT06350175
Title: Emergency Department Based Management of Tobacco Use Disorder
Brief Title: Emergency Department Management of Tobacco Use Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of participant/departmental interest. Nearing end of pilot grant award.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Bradley End, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2212697123
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-01-02 (Actual); Status verified 2024-12

CONDITIONS: Tobacco Use Disorder; Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotine Replacement Therapy (NRT) (Active Comparator): Subject provided with a 2-week supply of NRT and a West Virginia Quit Line (WV QL) fact sheet/contact information.
  Interventions: Combination Product: Nicotine Replacement Therapy Agent; Other: West Virginia Quit Line
- Control Non NRT Therapy (Other): Subject will be provided with a box/bag containing a WV QL fact sheet/contact information.
  Interventions: Other: West Virginia Quit Line

INTERVENTIONS:
Combination Product: Nicotine Replacement Therapy Agent — The NRT Agents-- 21mg nicotine patches (x14) and 2 mg nicotine lozenges (~210).
  Arms: Nicotine Replacement Therapy (NRT)
Other: West Virginia Quit Line — Instructional Pamphlets and contact information for the WV QL. A telehealth line set up to assist people of WV to quit smoking.

SUMMARY:
The objective of this study is to determine the effectiveness of ED initiated NRT on tobacco cessation point abstinence rates as reported by patients at 2 weeks and 1 month post randomization, and continued abstinence rates at 3 months compared to standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Current daily use cigarettes greater than or equal to ½ pack per day
* Stable for discharge from the ED
* Able and willing to complete telephone/electronic follow up at scheduled intervals
* Reported English speaking

Exclusion Criteria:

* Patients enrolled in specific health insurance plans (PEIA, The Health Plan or Medicaid medical insurance)
* WVU students
* Medically unstable patients
* Patients with clinical decompensation or who are admitted to the hospital
* Patients who are discharged to residential treatment facilities for detoxification
* Uncontrolled psychiatric disorder or psychiatric emergency
* Individuals who are unable to provide consent
* Incarcerated individuals
* Language barrier
* Currently pregnant or attempting to become pregnant
* Presenting for evaluation of sexual assault
* Known allergy or previous intolerance to nicotine replacement therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Continued Abstinence Rate (2 weeks) | 2 Weeks post initial dose
  Percentage of subjects who self-report continued abstinence in tobacco use at 2 weeks from initial dose given during the ED visit.
Percentage of Continued Abstinence Rate (1 month) | 1 Month post initial dose
  Percentage of subjects who self-report continued abstinence in tobacco use at 1 month from initial dose given during the ED visit.
Percentage of Continued Abstinence Rate (3 months) | 3 Months post initial dose
  Percentage of subjects who self-report continued abstinence in tobacco use at 3 months from initial dose given during the ED visit.
Patient Health Questionnaire 2 (Baseline) | Baseline
  A validated instrument to assess the frequency of depression and anhedonia screen for depression, scores can range from 0 to 6, with each item scored from 0 (not at all) to 3 (nearly every day). Scores greater than or equal to typically indicate depression.
Patient Health Questionnaire 2 (3 months from baseline) | 3 months from baseline
  A validated instrument to assess the frequency of depression and anhedonia screen for depression, scores can range from 0 to 6, with each item scored from 0 (not at all) to 3 (nearly every day). Scores greater than or equal to typically indicate depression.
Heaviness of Smoking Index (Baseline) | Baseline
  A validated measure used to determine the level of nicotine addiction, with a scale of 0-6 (3 indicates moderate addiction, >5 is severe)
Heaviness of Smoking Index (3 months from baseline) | 3 months from baseline
  A validated measure used to determine the level of nicotine addiction, with a scale of 0-6 (3 indicates moderate addiction, >5 is severe)
Richmond Test (Baseline) | Baseline
  A validated instrument to assess motivation to quit smoking. This is scored on a 0-10 scale with 5-6 indicating moderate motivation to quit and 7+ indicating strong motivation to quit.
Richmond Test (3 months from baseline) | 3 months from baseline
  A validated instrument to assess motivation to quit smoking. This is scored on a 0-10 scale with 5-6 indicating moderate motivation to quit and 7+ indicating strong motivation to quit.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley End, Principal Investigator — West Virginia University